CLINICAL TRIAL: NCT01621009
Title: A Randomized Controlled Clinical Trial of Bupropion SR and Individual Smoking Cessation Counseling
Brief Title: Bupropion SR Plus Counseling for Smoking Cessation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1998-369; P50CA084724 (NIH); P50DA019706 (NIH)
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: Tobacco Dependence; Smoking
Keywords: smoking cessation medications; smoking cessation counseling
MeSH Terms: conditions — Tobacco Use Disorder; Smoking | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (4):
- Active bupropion + counseling (Active Comparator): Active bupropion SR plus eight 10-minute individual counseling sessions.
  Interventions: Drug: Active bupropion + counseling
- Active bupropion , No counseling (Active Comparator): Active bupropion, No counseling, only medication checks
  Interventions: Drug: Active bupropion, No counseling
- Placebo medication + counseling (Placebo Comparator): Placebo bupropion plus eight 10-minute individual counseling sessions
  Interventions: Drug: Placebo medication + counseling
- Placebo medication, No counseling (Placebo Comparator): Placebo bupropion, No counseling, just medication checks
  Interventions: Drug: Placebo medication, No counseling

INTERVENTIONS:
Drug: Active bupropion + counseling — Medications-Pre-quit: 150 mg bupropion per day 7 days before quit attempt, then 150 mg twice daily for 4 days before quit attempt; then 150 mg bupropion twice daily for eight weeks.
  Counseling-Pre-quit: two 10 minutes sessions before quit date; eight 10-minute sessions post quit date.
  Arms: Active bupropion + counseling
Drug: Active bupropion, No counseling — Medication - 150 mg bupropion per day starting week before quit day, then 150 mg twice daily 3 days before quit day, then 150 mg twice daily for eight weeks after quit day.
  Counseling: No cessation counseling, only medication checks
  Arms: Active bupropion , No counseling
Drug: Placebo medication + counseling — Placebo bupropion once daily 7 days before quit day, then twice daily 4 days before quit attempt, then twice daily for 8 weeks after quit day.
  Counseling: Two 10-minutes sessions before quit day, then eight 10-minutes sessions for eight weeks after quit day.
  Arms: Placebo medication + counseling
Drug: Placebo medication, No counseling — Pre-quit: Placebo medication once daily 7 days before quit day, then twice daily before quit day, then twice daily for 8 weeks after quit day.
  Counseling: No counseling, just medication checks
  Arms: Placebo medication, No counseling

SUMMARY:
The purpose of this study was to determine if bupropion plus counseling was more effective than bupropion alone or counseling alone in helping smokers quit smoking.

ELIGIBILITY:
Inclusion Criteria:

* Smoke 10 or more cigarettes per day
* Expired carbon monoxide (CO) level greater than 9 parts per million (ppm)
* Motivated to quit smoking (score of 3 on 4-point self-report scale)
* Willing to fulfill study requirements

Exclusion Criteria:

* Carbon monoxide breath test score below 9 ppm
* Serious psychopathology (bipolar disorder, psychosis)
* Center for Epidemiologic Studies Depression Scale CES-D)score over 16
* Contraindications for use of bupropion
* History of seizure disorder
* History of eating disorder
* Current heavy drinking
* Risk of pregnancy
* Current breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 463 (Actual)
Dates: Start 2001-01; Primary Completion 2002-10 (Actual); Study Completion 2003-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy B Baker, PhD, Principal Investigator — University of Wisconsin, Madison; Timothy B Baker, PhD, Study Director — University of Wisconsin, Madison
Locations (1):
- UW Center for Tobacco Research and Intervention, Madison, Wisconsin, United States

REFERENCES:
- [Result] McCarthy DE, Piasecki TM, Lawrence DL, Jorenby DE, Shiffman S, Fiore MC, Baker TB. A randomized controlled clinical trial of bupropion SR and individual smoking cessation counseling. Nicotine Tob Res. 2008 Apr;10(4):717-29. doi: 10.1080/14622200801968343. PMID 18418793
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from Madison, WI area through TV, radio, newspaper advertisements from January, 2001 to October 2002
Pre-assignment Details: Participants were 1) phone screened, 2) invited to group orientation where signed consent was obtained, and 3) completed CO testing and office visit for physical exam. Participants were considered enrolled after passing all 3 steps and randomization occurred at enrollment.
Period: Overall Study
Arm/Group | Active Bupropion + Counseling | Active Bupropion , No Counseling | Placebo Medication + Counseling | Placebo Medication, No Counseling
Started | 113 | 116 | 121 | 113
Completed | 70 | 65 | 58 | 60
Not Completed | 43 | 51 | 63 | 53

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Bupropion + Counseling | Active Bupropion , No Counseling | Placebo Medication + Counseling | Placebo Medication, No Counseling | Total
Number analyzed (Participants) | 113 | 116 | 121 | 113 | 463
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 113 | 116 | 121 | 113 | 463
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.76 (11.39) | 41.03 (12.64) | 37.82 (12.82) | 39.42 (11.34) | 38.76 (12.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 57 | 63 | 61 | 233
  Male | 61 | 59 | 58 | 52 | 230
Region of Enrollment [Number; unit: participants]
  United States | 113 | 116 | 121 | 113 | 463
7-day point prevalence abstinence [Number; unit: participants] — Participants provided breath samples for carbon monoxide(CO)testing at all visits and provided a blood sample to assess cotinine (the first metabolite of nicotine)levels at baseline and again at end of treatment.
  participants
    Abstinent | 21 | 16 | 15 | 14 | 66
    Not Abstinent | 92 | 100 | 106 | 99 | 397

OUTCOME MEASURES:

1. Primary Outcome: 7-day Point Prevalence Abstinence From Smoking at 6 Months
Description: No smoking, not even a puff, during the 7 days prior to the 6 month follow-up. Biochemically confirmed.
Time Frame: 6 months
Population: Full intent-to-treat sample
Measure: Number; unit: Number of abstinent participants
Groups:
- Bupropion + Counseling: Active bupropion + 8 weeks counseling: Medications: Pre-quit - 150mg bupropion SR per day 3 days before quit day, then 150mg twice a day 4 days before quit day; 150mg bupropion SR twice daily for 8 weeks after the quit date.
  Counseling: Pre-quit - Two 10-minute sessions; Post-quit: Eight weekly 10-minute sessions
- Bupropion, No Counseling: Active bupropion, No counseling: Medications: Medications: Pre-quit - 150mg bupropion SR per day 3 days before quit day, then 150mg twice a day 4 days before quit day; 150mg bupropion SR twice daily for 8 weeks after the quit date. No cessation counseling, medication management and assessment only.
- Placebo + Counseling: : Medications: Pre-quit - Placebo bupropion one per day 3 days before quit day, then two per day 4 days before quit day; placebo bupropion twice daily for 8 weeks after the quit date.
  Counseling: Pre-quit - Two 10-minute sessions; Post-quit: Eight weekly 10-minute sessions
- Placebo, No Counseling: : Medications: Pre-quit - Placebo bupropion one per day 3 days before quit day, then two per day 4 days before quit day; placebo bupropion twice daily for 8 weeks after the quit date.
  No cessation counseling, medication management and assessment only.
Arm/Group | Bupropion + Counseling | Bupropion, No Counseling | Placebo + Counseling | Placebo, No Counseling
Number analyzed (Participants) | 113 | 116 | 121 | 113
Number of abstinent participants | 21 | 16 | 15 | 14
Statistical Analysis 1: Comparison: Bupropion + Counseling vs Placebo, No Counseling; Test type: Superiority or Other; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 1.61, 95% CI 2-sided [.78 to 3.36]
Statistical Analysis 2: Comparison: Bupropion + Counseling vs Bupropion, No Counseling; Test type: Superiority or Other; p > 0.05, Regression, Logistic; Odds Ratio (OR) = 1.13, 95% CI 2-sided [.52 to 2.44]

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Placebo Medication: Medications: Pre-quit - one placebo pill for 3 days before quit day, then one placebo pill twice a day 4 days before quit day for 8 weeks after the quit date.
- Active Medication: Pre-quit - 150mg bupropion SR per day 3 days before quit day, then 150mg twice a day 4 days before quit day; 150mg bupropion SR twice daily for 8 weeks after the quit date.
Arm/Group | Placebo Medication | Active Medication
Serious Adverse Events (participants affected / at risk) | 0/234 | 0/229
Other Adverse Events (participants affected / at risk) | 66/234 | 94/229
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Medication (N=234) | Active Medication (N=229)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 21 (21) | 19 (19)
depression (Nervous system disorders) | 25 (25) | 15 (15)
insomnia (Nervous system disorders) | 10 (10) | 35 (35)
Headache (Nervous system disorders) | 5 (5) | 14 (14)
Feeling jittery (Psychiatric disorders) | 5 (5) | 11 (11)

LIMITATIONS AND CAVEATS:
Lack of a no-treatment control condition; limited ability to generalize to broader population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes